CLINICAL TRIAL: NCT01358981
Title: Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single Escalating Oral Doses of LY2881835 in Healthy Subjects and Patients With Type 2 Diabetes Mellitus
Brief Title: A Study of LY2881835 in Healthy People and People With Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 13747; I4P-FW-GPFA (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-05-20; First posted 2011-05-24 (Estimated); Results first posted 2019-06-19 (Actual); Last update posted 2019-06-19 (Actual); Status verified 2019-03

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — LY2881835

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- LY2881835 (Experimental): One cohort of healthy participants will receive single oral doses of LY2881835 in up to 3 of the 4 periods in Part A (dose escalation: 0.5 milligram (mg), 1.5 mg, subsequent doses determined based on review of safety, tolerability, glycaemic response and available pharmacokinetic (PK) data from the first 2 dose levels). One cohort of participants with Type 2 Diabetes Mellitus (T2DM) will receive single oral doses of LY2881835 in up to 2 of the 3 periods in Part B (dose escalation: starting dose based on review of safety, tolerability, glycaemic response and available PK data from Part A).
  There is a washout period of at least 5 days between periods (doses).
  Interventions: Drug: LY2881835
- placebo (Placebo Comparator): One cohort of healthy participants will receive a single oral dose of placebo in 1 of the 4 periods in Part A. Another cohort of participants with T2DM will receive a single oral dose of placebo in 1 of the 3 periods in Part B.
  There is a washout period of at least 5 days between periods (doses).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY2881835 — Administered orally
  Arms: LY2881835
Drug: Placebo — Administered orally
  Arms: placebo

SUMMARY:
This will be the first study in which LY2881835 is given to humans in order to evaluate the safety and any side effects of LY2881835 in humans as well as how long LY2881835 stays in the body and its effect on blood sugar levels.

The study consists of two parts. In part A, healthy subjects will participate and in part B, patients with type 2 Diabetes Mellitus (T2DM) will participate.

ELIGIBILITY:
Inclusion Criteria:

All subjects:

* Are a healthy male or a healthy female who cannot become pregnant, or are patients with Type 2 Diabetes Mellitus (T2DM) who are not taking any drugs to lower blood sugar except metformin
* Have a body mass index (BMI) of at least 18.5 kilograms per meter squared (kg/m²) at screening
* Have blood pressure, pulse rate and clinical laboratory tests within the normal range for the population or investigator site, or with abnormalities deemed clinical insignificant by the investigator
* Have veins that are suitable for easy blood collection
* Are reliable and willing to be available for the whole study and are willing to follow study procedures
* Must have given written informed consent

Subjects with Type 2 Diabetes Mellitus (T2DM) only:

* Do not have any change to their diabetes treatment for at least 4 weeks prior to screening
* Have a glycosylated hemoglobin (HbA1c) level greater than or equal to 6% and less than or equal to 11% at screening

Exclusion Criteria:

All subjects:

* Are currently participating in or were in another new drug or medical research study in the last 30 days
* Have participated in this study before
* Have known allergies to compounds related to the study drug
* Currently have or used to have health problems or laboratory test results that in the opinion of the doctor, could interfere with understanding the results of this study
* Intend to use over-the-counter or prescription medications within 14 days prior to dosing or during the study. Hormone replacement therapy and intermittent use of paracetamol during the study is acceptable. For patients with Type 2 Diabetes Mellitus, medicines for control of high fats (For example, cholesterol), high blood pressure, are allowed.
* Have electrocardiogram (ECG) readings that are not suitable for the study
* Are unwilling to follow dietary restrictions/requirements for the study including 1) refrain from consuming foods or beverages containing grapefruit pomelo, star fruit, or Seville orange within 14 days of the start of the study drug dosing until collection of the last blood sample for drug assay and 2) consume only the meals provided during inpatient stays at the clinical research unit
* Have a history of drug or alcohol abuse
* Are infected with hepatitis B
* Are infected with human immunodeficiency disease virus (HIV)
* Have donated 450 milliliters (mL) or more of blood in the last 3 months or provided any blood donation within the last month from screening
* Have a regular alcohol intake greater than 21 units per week (males) and 14 units per week (females) or are not willing to abstain from alcohol while in the research unit
* Smoke more than 10 cigarettes per day or are not willing to abstain from smoking while at the clinic
* The study doctor thinks the subject should not participate for any other reasons

Subjects with Type 2 Diabetes Mellitus (T2DM) only:

* Have health complications due to poorly controlled diabetes as shown by blood and urine laboratory test results or based on physical examination and medical assessment, as determined by the study doctor
* Were hospitalised for poor control of their diabetes (ketoacidotic episode) in the last 6 months
* Currently using or have used insulin in the last 1 year to control their diabetes

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-05-24 (Actual); Primary Completion 2011-08-17 (Actual); Study Completion 2011-08-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Yes
Lilly provides access to the individual patient data from studies on approved medicines and indications as defined by the sponsor specific information on ClinicalStudyDataRequest.com.
  This access is provided in a timely fashion after the primary publication is accepted. Researchers need to have an approved research proposal submitted through ClinicalStudyDataRequest.com. Access to the data will be provided in a secure data sharing environment after signing a data sharing agreement.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is a 2-part (Part A and Part B) crossover study with four periods.In Part A, 8 participants were dosed at each dose level in 4 study periods (1 additional participant was dosed only in 1 study period). In Part B, a single cohort of 9 participants with type 2 diabetes mellitus (T2DM) participated in 3 dosing periods.
Groups:
- Cohort 1: Part A (Healthy): Sequence 1: Participants received single oral doses of 0.5 milligram (mg), 1.5 mg, 4.5 mg LY2881835 and placebo capsules on day 1 of each treatment period as per the below dosing sequence.
  Period 1: 0.5 mg LY2881835, Period 2: 1.5 mg LY2881835, Period 3: 4.5 mg LY2881835, Period 4: Placebo.
- Cohort 1: Part A (Healthy): Sequence 2: Participants received single oral doses of 0.5 mg, 1.5 mg, 8.4 mg LY2881835 and placebo capsules on day 1 of each treatment period as per the below dosing sequence.
  Period 1: 0.5 mg LY2881835, Period 2: 1.5 mg LY2881835, Period 3: Placebo, Period 4: 8.4 mg LY2881835.
- Cohort 1: Part A (Healthy): Sequence 3: Participants received single oral doses of 0.5 mg, 4.5 mg, 8.4 mg LY2881835 and placebo capsules on day 1 of each treatment period as per the below dosing sequence.
  Period 1: 0.5 mg LY2881835, Period 2: Placebo, Period 3: 4.5 mg LY2881835, Period 4: 8.4 mg LY2881835.
- Cohort 1: Part A (Healthy): Sequence 4: Participants received single oral doses of 1.5 mg, 4.5 mg, 8.4 mg LY2881835 and placebo capsules on day 1 of each treatment period as per the below dosing sequence.
  Period 1: Placebo, Period 2: 1.5 mg LY2881835, Period 3: 4.5 mg LY2881835, Period 4: 8.4 mg LY2881835.
- Cohort 2: Part B (T2DM): Sequence 1: Participants received single oral doses of 8.4 mg LY2881835 and placebo capsules on day 1 of each treatment period as per the below dosing sequence.
  Period 1: 8.4 mg LY2881835, Period 2: 8.4 mg LY2881835, Period 3: Placebo.
- Cohort 2: Part B (T2DM): Sequence 2: Participants received single oral doses of 8.4 mg LY2881835 and placebo capsules on day 1 of each treatment period as per the below dosing sequence.
  Period 1: 8.4 mg LY2881835, Period 2: Placebo, Period 3: 8.4 mg LY2881835.
- Cohort 2: Part B (T2DM): Sequence 3: Participants received single oral doses of 8.4 mg LY2881835 and placebo capsules on day 1 of each treatment period as per the below dosing sequence.
  Period 1: Placebo, Period 2: 8.4 mg LY2881835, Period 3: 8.4 mg LY2881835.
Period: Period 1
Arm/Group | Cohort 1: Part A (Healthy): Sequence 1 | Cohort 1: Part A (Healthy): Sequence 2 | Cohort 1: Part A (Healthy): Sequence 3 | Cohort 1: Part A (Healthy): Sequence 4 | Cohort 2: Part B (T2DM): Sequence 1 | Cohort 2: Part B (T2DM): Sequence 2 | Cohort 2: Part B (T2DM): Sequence 3
Started | 2 | 2 | 2 | 2 | 3 | 3 | 3
Received at Least 1dose of Study Drug | 2 | 2 | 2 | 2 | 3 | 3 | 3
Completed | 2 | 2 | 2 | 1 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0 | 0
Period: Period 2
Arm/Group | Cohort 1: Part A (Healthy): Sequence 1 | Cohort 1: Part A (Healthy): Sequence 2 | Cohort 1: Part A (Healthy): Sequence 3 | Cohort 1: Part A (Healthy): Sequence 4 | Cohort 2: Part B (T2DM): Sequence 1 | Cohort 2: Part B (T2DM): Sequence 2 | Cohort 2: Part B (T2DM): Sequence 3
Started | 2 | 2 | 2 | 2 (One participant who withdrew in period 1 was replaced by another participant in period 2.) | 3 | 3 | 3
Completed | 2 | 2 | 2 | 2 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Cohort 1: Part A (Healthy): Sequence 1 | Cohort 1: Part A (Healthy): Sequence 2 | Cohort 1: Part A (Healthy): Sequence 3 | Cohort 1: Part A (Healthy): Sequence 4 | Cohort 2: Part B (T2DM): Sequence 1 | Cohort 2: Part B (T2DM): Sequence 2 | Cohort 2: Part B (T2DM): Sequence 3
Started | 2 | 2 | 2 | 2 | 3 | 3 | 3
Completed | 2 | 2 | 2 | 2 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 4
Arm/Group | Cohort 1: Part A (Healthy): Sequence 1 | Cohort 1: Part A (Healthy): Sequence 2 | Cohort 1: Part A (Healthy): Sequence 3 | Cohort 1: Part A (Healthy): Sequence 4 | Cohort 2: Part B (T2DM): Sequence 1 | Cohort 2: Part B (T2DM): Sequence 2 | Cohort 2: Part B (T2DM): Sequence 3
Started | 2 | 2 | 2 | 2 | 0 (Part B was planned for only 3 dosing periods.) | 0 (Part B was planned for only 3 dosing periods.) | 0 (Part B was planned for only 3 dosing periods.)
Completed | 2 | 2 | 2 | 2 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Part A (Healthy): Sequence 1 | Cohort 1: Part A (Healthy): Sequence 2 | Cohort 1: Part A (Healthy): Sequence 3 | Cohort 1: Part A (Healthy): Sequence 4 | Cohort 2: Part B (T2DM): Sequence 1 | Cohort 2: Part B (T2DM): Sequence 2 | Cohort 2: Part B (T2DM): Sequence 3 | Total
Number analyzed (Participants) | 2 | 2 | 2 | 3 | 3 | 3 | 3 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 2 | 3 | 3 | 3 | 3 | 18
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 1 | 0 | 2 | 2 | 3 | 8
  Male | 2 | 2 | 1 | 3 | 1 | 1 | 0 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 2 | 2 | 3 | 3 | 3 | 3 | 18
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 2 | 2 | 3 | 3 | 3 | 3 | 18
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Singapore | 2 | 2 | 2 | 3 | 3 | 3 | 3 | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinically Significant Adverse Effects
Description: Clinically significant adverse effects are treatment emergent adverse events (TEAEs) possibly related to study drug.
Time Frame: Baseline to study completion up to 3 months
Population: All enrolled participants who received study drug.
Measure: Number; unit: participants
Groups:
- Part A - Placebo: Single oral dose of placebo in a study period in Part A (Healthy).
- Part A - 0.5 mg LY2881835: Single oral dose of 0.5 milligram (mg) LY2881835 in a study period in Part A (Healthy).
- Part A - 1.5 mg LY2881835: Single oral dose of 1.5 mg LY2881835 in a study period in Part A (Healthy).
- Part A - 4.5 mg LY2881835: Single oral dose of 4.5 mg LY2881835 in a study period in Part A (Healthy).
- Part A - 8.4 mg LY2881835: Single oral dose of 8.4 mg LY2881835 in a study period in Part A (Healthy).
- Part B - Placebo: Single oral dose of placebo in a study period in Part B [Type 2 Diabetes Mellitus (T2DM)].
- Part B - 8.4 mg LY2881835: Single oral dose of 8.4 mg LY2881835 in 2 of the 3 study periods in Part B (T2DM).
Arm/Group | Part A - Placebo | Part A - 0.5 mg LY2881835 | Part A - 1.5 mg LY2881835 | Part A - 4.5 mg LY2881835 | Part A - 8.4 mg LY2881835 | Part B - Placebo | Part B - 8.4 mg LY2881835
Number analyzed (Participants) | 9 | 6 | 6 | 6 | 6 | 9 | 9
participants | 0 | 0 | 1 | 0 | 0 | 1 | 2

2. Secondary Outcome: Pharmacokinetics (PK): Area Under the Curve (AUC) of LY2881835
Description: Not all the participants had quantifiable plasma concentrations at 48 hours, therefore only AUC from time zero to 24 hours [AUC(0-24 hours)] is provided.
Time Frame: Part A: Predose, 0.5, 1.5, 2.5, 4, 6, 12, 18 and 24hours (h) post-dose; Part B: Predose, 0.5, 1.5, 2.5, 4, 6, 12, 18 and 24 h post-dose
Population: All participants who received study drug and had evaluable PK data. Each participant in group Part B, Study Periods 1, 2 and 3 - 8.4 mg LY2881835 was dosed and had corresponding PK measures in 2 of the 3 study periods in Part B resulting in 18 samples being analyzed. Analysis used data according to the treatment the participants actually received.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour/milliliter (ng*hr/mL)
Units Other Than Participants: Samples
Groups:
- Part B, Study Period 1 - 8.4 mg LY2881835: Single oral dose of 8.4 mg LY2881835 in Study Period 1 in Part B [Type 2 Diabetes Mellitus (T2DM)].
- Part B, Study Period 2 - 8.4 mg LY2881835: Single oral dose of 8.4 mg LY2881835 in Study Period 2 in Part B (T2DM).
- Part B, Study Period 3 - 8.4 mg LY2881835: Single oral dose of 8.4 mg LY2881835 in Study Period 3 in Part B (T2DM).
- Part B, Study Periods 1, 2, and 3 - 8.4 mg LY2881835: Single oral dose of 8.4 mg LY2881835 in 2 of the 3 study periods in Part B (T2DM).
Arm/Group | Part A - 0.5 mg LY2881835 | Part A - 1.5 mg LY2881835 | Part A - 4.5 mg LY2881835 | Part A - 8.4 mg LY2881835 | Part B, Study Period 1 - 8.4 mg LY2881835 | Part B, Study Period 2 - 8.4 mg LY2881835 | Part B, Study Period 3 - 8.4 mg LY2881835 | Part B, Study Periods 1, 2, and 3 - 8.4 mg LY2881835
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 9
Number analyzed (Samples) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 18
nanograms*hour/milliliter (ng*hr/mL) | 54.8 (39) | 125 (47) | 340 (31) | 767 (48) | 820 (20) | 683 (26) | 658 (43) | 717 (31)

3. Secondary Outcome: Pharmacokinetics (PK): Maximum Concentration (Cmax) Of LY2881835
Description: Not all the participants had quantifiable plasma concentrations at 48 hours, therefore only Cmax up to 24 hours post-dose is provided.
Time Frame: Part A: Predose, 0.5, 1.5, 2.5, 4, 6, 12, 18 and 24 h post-dose; Part B: Predose, 0.5, 1.5, 2.5, 4, 6, 12, 18 and 24 h post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliter (ng/mL)
Units Other Than Participants: Samples
Arm/Group | Part A - 0.5 mg LY2881835 | Part A - 1.5 mg LY2881835 | Part A - 4.5 mg LY2881835 | Part A - 8.4 mg LY2881835 | Part B, Study Period 1 - 8.4 mg LY2881835 | Part B, Study Period 2 - 8.4 mg LY2881835 | Part B, Study Period 3 - 8.4 mg LY2881835 | Part B, Study Periods 1, 2, and 3 - 8.4 mg LY2881835
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 9
Number analyzed (Samples) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 18
nanograms/milliliter (ng/mL) | 7.44 (16) | 14.7 (38) | 47.1 (25) | 89.9 (42) | 93.0 (30) | 85.1 (32) | 77.8 (21) | 85.1 (27)

4. Secondary Outcome: Pharmacokinetics (PK): Time to Maximum Concentration (Tmax) of LY2881835
Description: Not all the participants had quantifiable plasma concentrations at 48 hours, therefore only Tmax up to 24 hours post dose is provided.
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Units Other Than Participants: Samples
Arm/Group | Part A - 0.5 mg LY2881835 | Part A - 1.5 mg LY2881835 | Part A - 4.5 mg LY2881835 | Part A - 8.4 mg LY2881835 | Part B, Study Period 1 - 8.4 mg LY2881835 | Part B, Study Period 2 - 8.4 mg LY2881835 | Part B, Study Period 3 - 8.4 mg LY2881835 | Part B, Study Periods 1, 2, and 3 - 8.4 mg LY2881835
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 18
Number analyzed (Samples) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 18
hours | 2.50 [1.50 to 4.00] | 2.50 [1.50 to 4.00] | 3.25 [2.50 to 6.00] | 2.50 [1.50 to 4.02] | 4.25 [1.50 to 6.00] | 3.25 [2.50 to 6.00] | 4.25 [1.50 to 6.00] | 3.25 [1.50 to 6.00]

5. Secondary Outcome: Glucose Area Under the Effective Concentration Curve (AUEC)
Description: Glucose area under the serum concentration versus time curve (AUEC) was calculated using the linear trapezoidal rule from time 0 to 24 hours.
Time Frame: Part A: Predose, 1.0, 1.5, 2.5, 3.5, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 18 and 24 h post-dose; Part B: Predose, 1.0, 1.5, 2.5, 3.5, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 18 and 24 h post-dose
Population: All participants who received study drug and had evaluable glucose data. Each participant in group Part B, Study Periods (SP) 1, 2 and 3-8.4 mg LY2881835 was dosed and had corresponding glucose measures in 2 of the 3 SP in Part B resulting in 18 samples being analyzed. Analysis used data according to the treatment participants actually received.
Measure: Mean (Standard Deviation); unit: milligrams*hour/deciliter (mg*hr/dL)
Units Other Than Participants: Samples
Arm/Group | Part A - Placebo | Part A - 0.5 mg LY2881835 | Part A - 1.5 mg LY2881835 | Part A - 4.5 mg LY2881835 | Part A - 8.4 mg LY2881835 | Part B - Placebo | Part B - 8.4 mg LY2881835
Number analyzed (Participants) | 9 | 6 | 6 | 6 | 6 | 9 | 9
Number analyzed (Samples) | 9 | 6 | 6 | 6 | 6 | 9 | 18
milligrams*hour/deciliter (mg*hr/dL) | 2282 (291) | 2448 (183) | 2089 (146) | 2354 (72) | 2159 (133) | 3640 (711) | 3769 (719)

6. Secondary Outcome: Glucagon-Like Peptide (Active GLP-1) Area Under the Effective Concentration Curve (AUEC)
Description: Glucagon-like peptide (active GLP-1) area under the serum concentration versus time curve (AUEC) was calculated using the linear trapezoidal rule from time 0 to 2.5 hours.
Time Frame: Part A: Predose, 1.5 and 2.5 h post-dose; Part B: Predose, 1.5 and 2.5 h post-dose
Population: All participants who received study drug and had evaluable GLP-1 data. Each participant in group Part B, Study Periods (SP) 1, 2 and 3-8.4 mg LY2881835 was dosed and had corresponding GLP-1 measures in 2 of the 3 SP in Part B resulting in 18 samples being analyzed. Analysis used data according to the treatment participants actually received.
Measure: Mean (Standard Deviation); unit: picomoles*hour/liter (pmol*h/L)
Units Other Than Participants: Samples
Groups:
- Part A - 0.5 mg LY2881835: Single oral dose of 0.5 mg LY2881835 in a study period in Part A (Healthy).
Arm/Group | Part A - Placebo | Part A - 0.5 mg LY2881835 | Part A - 1.5 mg LY2881835 | Part A - 4.5 mg LY2881835 | Part A - 8.4 mg LY2881835 | Part B - Placebo | Part B - 8.4 mg LY2881835
Number analyzed (Participants) | 9 | 6 | 6 | 6 | 6 | 9 | 9
Number analyzed (Samples) | 9 | 6 | 6 | 6 | 6 | 9 | 18
picomoles*hour/liter (pmol*h/L) | 3.029 (1.097) | 3.277 (1.032) | 2.838 (0.759) | 3.113 (1.389) | 3.362 (0.938) | 4.249 (2.140) | 5.268 (2.266)

7. Secondary Outcome: C-Peptide Area Under the Effective Concentration Curve (AUEC)
Description: C-Peptide area under the serum concentration versus time curve (AUEC) was calculated using the linear trapezoidal rule from time 0 to 6 hours.
Time Frame: Part A: Predose, 1.0, 1.5, 2.5, 4, 5, 6 and 24 h post-dose; Part B: Predose, 1.0, 1.5, 2.5, 4, 5, 6 and 24 h post-dose
Population: All participants who received study drug and had evaluable C-Peptide data. Each participant in group Part B, Study Periods (SP) 1, 2, 3-8.4 mg LY2881835 was dosed and had corresponding C-Peptide measures in 2 of the 3 SP in Part B resulting in 18 samples being analyzed. Analysis used data according to the treatment participants actually received.
Measure: Mean (Standard Deviation); unit: picomoles*hour/liter (pmol*h/L)
Units Other Than Participants: Samples
Arm/Group | Part A - Placebo | Part A - 0.5 mg LY2881835 | Part A - 1.5 mg LY2881835 | Part A - 4.5 mg LY2881835 | Part A - 8.4 mg LY2881835 | Part B - Placebo | Part B - 8.4 mg LY2881835
Number analyzed (Participants) | 9 | 6 | 6 | 6 | 6 | 9 | 9
Number analyzed (Samples) | 9 | 6 | 6 | 6 | 6 | 9 | 18
picomoles*hour/liter (pmol*h/L) | 5852.8 (1266.7) | 6313.7 (1870.3) | 7069.5 (2065.3) | 4962.2 (1192.2) | 7421.5 (3047.4) | 6145.6 (2192.4) | 6477.8 (2113.4)

ADVERSE EVENTS:
Time Frame: Baseline to study completion up to 3 months
Description: All enrolled participants who received study drug.
Arm/Group | Part A - Placebo | Part A - 0.5 mg LY2881835 | Part A - 1.5 mg LY2881835 | Part A - 4.5 mg LY2881835 | Part A - 8.4 mg LY2881835 | Part B - Placebo | Part B - 8.4 mg LY2881835
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/6 | 0/6 | 0/6 | 0/6 | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/6 | 0/6 | 0/6 | 0/6 | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 3/9 | 3/6 | 3/6 | 2/6 | 4/6 | 3/9 | 4/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A - Placebo (N=9) | Part A - 0.5 mg LY2881835 (N=6) | Part A - 1.5 mg LY2881835 (N=6) | Part A - 4.5 mg LY2881835 (N=6) | Part A - 8.4 mg LY2881835 (N=6) | Part B - Placebo (N=9) | Part B - 8.4 mg LY2881835 (N=9)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Catheter site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Catheter site pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hunger (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Vessel puncture site swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural site reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No